CLINICAL TRIAL: NCT03697408
Title: An Open-Label Phase I/II Safety and Efficacy Study of Itacitinib In Combination With Everolimus In Subjects With Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Itacitinib + Everolimus in Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 831774; UPCC #45418
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — itacitinib; INCB039110; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort -1 (Experimental): Itacitinib 200 mg once daily (QD) in combination with everolimus 5 mg QD
  Interventions: Drug: Itacitinib; Drug: Everolimus
- Cohort 1 (starting dose) (Experimental): Itacitinib 300 mg once daily (QD) in combination with everolimus 5 mg QD
  Interventions: Drug: Itacitinib; Drug: Everolimus
- Cohort 2 (Experimental): Itacitinib 400 mg once daily (QD) in combination with everolimus 5 mg QD
  Interventions: Drug: Itacitinib; Drug: Everolimus

INTERVENTIONS:
Drug: Itacitinib — A JAK 1 selective small molecule inhibitor
  Other Names: INCB039110
Drug: Everolimus — A mammalian target of rapamycin (mTOR) inhibitor
  Other Names: Afinitor

SUMMARY:
This is an open-label, single-group, Phase I/II study of itacitinib in combination with everolimus in subjects with relapsed or refractory classical Hodgkin lymphoma (cHL).

DETAILED DESCRIPTION:
This is an open-label, single-group, Phase I/II study of itacitinib in combination with everolimus in subjects with relapsed or refractory cHL. Phase I will evaluate the safety and tolerability of itacitinib when combined with everolimus in subjects with relapsed refractory cHL using a 3 + 3 design; Phase II will evaluate the efficacy of the combination in subjects with cHL at the dose determined in Phase I using a Simon 2-stage expansion design. Subjects may continue to receive study treatment for 2 years or until evidence of disease progression, unacceptable toxicity, inability to obtain commercial everolimus or consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the informed consent form.
2. Aged 18 years or older at the time of signing the informed consent form.
3. Biopsy-proven diagnosis of relapsed classical Hodgkin lymphoma.
4. Measurable disease on imaging defined as at least one lesion that can be accurately measured in at least two dimensions by imaging (PET/CT, CT or MRI). Minimum measurement must be ≥ 15mm in the longest axis or ≥ 10mm in the short axis.
5. Relapsed or refractory disease (after at least 2 prior systemic therapies); patients must have relapsed after high-dose therapy with ASCT, or have been deemed ineligible for high-dose therapy with ASCT based upon the below criteria:

   * Patients that have either progressed after treatment with, be intolerant to, or are not a candidate for brentuximab and pembrolizumab or nivolumab. The reason for forgoing such therapies must be clearly documented.
   * Are not ASCT candidates due to chemo-resistant disease (unable to achieve CR or PR to salvage chemotherapy), advanced age (≥ 65 years of age), or any significant coexisting medical condition (renal, pulmonary, or hepatic dysfunction) likely to have a negative impact on tolerability of ASCT
6. Disease free of other malignancies for greater than or equal to 2 years with the exception of basal cell, squamous cell carcinomas of the skin, fully excised melanoma in situ, carcinoma in situ of the cervix or breast.
7. Performance status of ECOG 0-2 (Appendix 13.3).
8. Laboratory test results within these ranges (of note, patients who have cytopenias due to documented cHL involvement of the bone marrow may be considered for enrollment after discussion with the PI, Medical Director and Sponsor):

   * Absolute neutrophil count (ANC) > 1,000/µL
   * Platelet count > 75,000/µL
   * Serum creatinine < 2.0 mg/dL
   * Bilirubin < 2.0 × ULN unless bilirubin increase was due to Gilbert's disease. Further evaluation should be performed to confirm and document the origin of increase.
   * AST and ALT ≤ 2.5 × institutional upper limit of normal (ULN)
   * Fasting cholesterol ≤ 300 mg/dL AND fasting triglycerides ≤ 300 mg/dl. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication prior initiating study treatment.
9. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 72 hours prior to the first dose of itacitinib and must agree to use an effective contraception method during the study and for 6 months following the last dose of study drug; females of non-childbearing potential are those who are post-menopausal for more than 1 year or who have had a bilateral tubal ligation or hysterectomy. Female patients undergoing active fertility preservation therapy/egg harvesting which include hCG injections are expected to have mild elevation of hCG. These patients may be allowed to participate in the trial despite elevation of hCG after providing documentation of negative hCG prior the hCG injection and statement from her fertility specialist that they are not pregnant.
10. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of study drug.
11. Must be able to comply with the study and follow-up requirements.
12. Subject must have access to everolimus via insurance or self-pay.

Exclusion Criteria:

1. Unable to sign informed consent form.
2. Pregnant or breast-feeding females (lactating females must agree not to breast feed while taking the investigational agents).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study. For Example:

   * symptomatic congestive heart failure of New York Heart Association Class III or IV
   * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   * severely impaired lung function with O2 saturation that is 88% or less at rest on room air
   * active (acute or chronic) or uncontrolled severe infections
   * condition requiring ongoing use of medications that are considered STRONG or MODERATE CYP3A4 inhibitors or inducers and P-gp substrates at study screening . However, those who require weak inhibitors/inducers can be enroll at discretion of the PI.
   * liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
4. Has a history (within the past 12 months) of (non-infectious) pneumonitis requiring systemic steroids, or active pneumonitis.
5. Bilirubin < 3 × ULN in the presence of liver metastases or presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia)
6. Concurrent use of other anti-cancer agents or therapies during study treatment.
7. Use of any other experimental drug or therapy within 28 days of initiating treatment with the investigational agents.
8. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis C (HCV), or hepatitis B virus (HBV); patients who are seropositive because of hepatitis B virus vaccine are eligible.
9. Previous use of JAK1 inhibitor (itacitinib), or history of progression on everolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2027-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Svoboda, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study: 23 evaluable subjects. Phase I: 6 to 15 subjects enrolled (with at least 6 subjects treated at the recommended Phase II dose (RP2D)). The itacitinib starting dose is 300 mg once daily (QD). Depending on tolerability, the itacitinib dose could be increased to 400 mg QD or decreased to 200 mg QD. The everolimus dose will remain 5 mg QD for each cohort.
  Phase II: Additional subjects will receive the RP2D of itacitinib with everolimus as determined in Phase I.
Period: Phase I (Dose Finding)
Arm/Group | Cohort 1 (Starting Dose) | Cohort -1 | Cohort 2
Started | 3 | 0 | 6
Completed | 3 | 0 | 6
Not Completed | 0 | 0 | 0
Period: Phase II (Treatment)
Arm/Group | Cohort 1 (Starting Dose) | Cohort -1 | Cohort 2
Started | 3 | 0 | 20 (14 additional subjects enrolled.)
Completed | 3 (One subject completed treatment at 200 mg itacitinib dose.) | 0 | 20 (Seven subjects completed treatment at the 300 mg itacitinib dose.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cohorts into which subjects with relapsed/refractory classical Hodgkin lymphoma (cHL) were enrolled. No subjects were enrolled into Cohort -1 (starting dose of itacitinib 200 mg in combination with everolimus 5 mg).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Starting Dose) | Cohort -1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 0 | 20 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 20 | 22
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 6 | 7
  Male | 2 | 0 | 14 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 0 | 19 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 4
  White | 3 | 0 | 16 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Efficacy of Itacitinib in Combination With Everolimus
Description: Evaluate the efficacy of itacitinib in combination with everolimus in subjects with relapsed or refractory cHL as demonstrated by complete response (CR) rate, defined as the percentage of subjects achieving CR as their best response.
Time Frame: 2 Years
Population: Efficacy will be assessed by CR rate, defined as the percentage of subjects achieving Complete Response (CR) as their best response
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving CR
Arm/Group | Cohort 1 (Starting Dose) | Cohort -1 | Cohort 2
Number analyzed (Participants) | 3 | 0 | 20
percentage of subjects achieving CR | 33.3 [10.2 to 90.5] |  | 25 [8.66 to 49.1]

2. Secondary Outcome: Determine the Efficacy of Itacitinib in Combination With Everolimus in Terms of Overall Response Rate (ORR).
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Determine the Efficacy of Itacitinib in Combination With Everolimus in Terms of Partial Response (PR).
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Determine the Efficacy of Itacitinib in Combination With Everolimus in Terms of Stable Disease (SD).
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Determine the Efficacy of Itacitinib in Combination With Everolimus in Terms of Duration of Response.
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Determine the Efficacy of Itacitinib in Combination With Everolimus in Terms of Progression Free Survival (PFS).
Time Frame: 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Determine the Efficacy of Itacitinib in Combination With Everolimus in Terms of Overall Survival (OS).
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data is collected from the time of informed consent until End-of-Treatment visit - 14 months
Description: Cohorts into which subjects with relapsed/refractory classical Hodgkin lymphoma (cHL) were enrolled. No subjects were enrolled into Cohort -1 (starting dose of itacitinib 200 mg in combination with everolimus 5 mg).
Arm/Group | Cohort 1 (Starting Dose) | Cohort -1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/0 | 7/20
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/0 | 6/20
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Starting Dose) (N=3) | Cohort -1 (N=0) | Cohort 2 (N=20)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Starting Dose) (N=3) | Cohort -1 (N=0) | Cohort 2 (N=20)
Anemia (Blood and lymphatic system disorders) | 3 (14) | 0 (0) | 18 (32)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 9 (9)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 6 (6)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 7 (13)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 10 (21)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Blood lactate dehydrogenase increased (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 17 (22)
Cholesterol high (Investigations) | 2 (3) | 0 (0) | 11 (13)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 7 (8)
Neutrophil count decreased (Investigations) | 1 (4) | 0 (0) | 9 (17)
Platelet count decreased (Investigations) | 2 (15) | 0 (0) | 18 (44)
White blood cell decreased (Investigations) | 2 (10) | 0 (0) | 13 (27)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 10 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 13 (13)
Hot flashes (Vascular disorders) | 2 (3) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (6) | 0 (0) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03697408/Prot_SAP_002.pdf
  • Informed Consent Form (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03697408/ICF_001.pdf